CLINICAL TRIAL: NCT06766149
Title: The Effects of Computerized Cognitive Training on Executive Function in Children in Hong Kong
Brief Title: CogniFit Computerized Cognitive Training in Primary School Students in Hong Kong
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Edge Development Centre (Unknown)
Responsible Party: Principal Investigator, Dr. Kathy Shum, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EA240316
Record Dates: First submitted 2025-01-03; First posted 2025-01-09 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Executive Function (Cognition)
Keywords: executive function; children; computerized cognitive training; working memory; cognitive function

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CogniFit Group (Experimental): The CogniFit training group will receive 24 sessions of training, 35 - 40 minutes each, conducted three times per week over a period of 8 weeks. Participants will be asked to complete a set of computerized tasks using CogniFit, a digital training programme which is proven to enhance cognitive ability of participants.
  Interventions: Behavioral: CogniFit Computerized Cognitive Training
- Cogmed Group (Active Comparator): The Cogmed training group will receive 24 sessions of training, 35 - 40 minutes each, conducted three times per week over a period of 8 weeks. Participants will be asked to complete a set of computerized tasks using Cogmed, a digital training programme which is proven to enhance working memory and attentional control of participants.
  Interventions: Behavioral: Cogmed Computerized Cognitive Training
- Waitlist Control Group (No Intervention): The waitlist control group will not receive any intervention until the intervention arms complete their training. After completion of the assessment at Timepoint 3, Computerized Cognitive Training will be offered to this group.

INTERVENTIONS:
Behavioral: CogniFit Computerized Cognitive Training — In the CogniFit Computerized Cognitive Training, children will complete a range of tasks covering a range of game-like exercises targeting various cognitive skills, including working memory, attention, and inhibitory control, with automatic level advancement after each exercise.
  Arms: CogniFit Group
Behavioral: Cogmed Computerized Cognitive Training — In the Cogmed Computerized Cognitive Training, children will complete a range of tasks covering a range of game-like exercises targeting various cognitive skills, including working memory and attentional control, with automatic level advancement after each exercise.
  Arms: Cogmed Group

SUMMARY:
This study aims to address these gaps by conducting a comprehensive evaluation of the effects of CogniFit training in children. The primary objective of this study is to evaluate the effectiveness of CogniFit training on executive functions among primary school students in Hong Kong.

Specific objectives include:

1. To assess the effectiveness of CogniFit training on improving executive functions, such as working memory, attention, and inhibitory control in children compared to a waitlist control group.
2. To assess the effectiveness of CogniFit training on improving executive functions, such as working memory, attention, and inhibitory control in children compared to an active control group that will receive Cogmed training.

Participants will be randomly assigned to one of three groups: 1) the CogniFit training group; 2) the Cogmed Group, and 3) the wailist controlled group.

Participants in the two computerized cognitive training groups (CogniFit/Cogmed Group) will receive training in the first phase of intervention, while the waitlist control group will CogniFit trainings in the second phase of intervention.

Participants who receive the computerized cognitive training will complete 24 sessions of training, 15-20 minutes each, conducted three times per week spanning 8 weeks. These programs comprise a range of game-like exercises targeting various cognitive skills, including working memory, attention, and inhibitory control, with automatic level advancement after each exercise.

To investigate the intervention effectiveness, children will be asked to complete a set of cognitive tests covering inhibitory control, attention, and working memory prior to the intervention (i.e., Time 1), immediately after the 8-week training (i.e., Time 2), and 2 months after the training (i.e., Time 3, a 2-month follow up). The assessment will take around 1 hour and it will be conducted at participants' schools. Also, parents will be asked to complete a questionnaire assessing children's behaviours at home and schools at 3 time points.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6- 12
* Studying in Grade 1 to 6 in mainstream primary schools in Hong Kong

Exclusion Criteria:

* Inability to answer the first five questions in Raven's Progressive Matrices
* Hearing, visual, or physical impairments that might hinder participation in the training and assessment activities
* Current participation in a computerized cognitive treatment

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Executive Functiong - Conners Continuous Performance Test 3rd Edition (CPT 3) | Pre-intervention Assessment (within 4 weeks before the commencement of the intervention)
  A standardized computerized test on sustained attention and inhibitory control
Executive Functiong - Conners Continuous Performance Test 3rd Edition (CPT 3) | Immediate Post-intervention Assessment (within 4 weeks after the completion of the intervention)
  A standardized computerized test on sustained attention and inhibitory control
Executive Functiong - Conners Continuous Performance Test 3rd Edition (CPT 3) | Delayed Post-intervention Assessment (a 2-month follow up after the completion of the intervention)
  A standardized computerized test on sustained attention and inhibitory control
Executive Function - Number subtest of Children's Memory Scale (CMS) | Pre-intervention Assessment (within 4 weeks before the commencement of the intervention)
  A verbal working memory test using digit span, with a higher score indicating a higher level of verbal working memory. The total score of this test ranges from 0 to 30.
Executive Function - Number subtest of Children's Memory Scale (CMS) | Immediate Post-intervention Assessment (within 4 weeks after the completion of the intervention)
  A verbal working memory test using digit span, with a higher score indicating a higher level of verbal working memory. The total score of this test ranges from 0 to 30.
Executive Function - Number subtest of Children's Memory Scale (CMS) | Delayed Post-intervention Assessment (a 2-month follow up after the completion of the intervention)
  A verbal working memory test using digit span, with a higher score indicating a higher level of verbal working memory. The total score of this test ranges from 0 to 30.

SECONDARY OUTCOMES:
Behavioural ratings on children's executive functions | Pre-intervention Assessment (within 4 weeks before the commencement of the intervention)
  Parents' report of Behavior Rating Inventory of Executive Function, Second Edition (BRIEF2) measuring a range of executive functions, including behavioural, emotional and cognitive regulation
Behavioural ratings on children's executive functions | Immediate Post-intervention Assessment (within 4 weeks after the completion of the intervention)
  Parents' report of Behavior Rating Inventory of Executive Function, Second Edition (BRIEF2) measuring a range of executive functions, including behavioural, emotional and cognitive regulation
Behavioural ratings on children's executive functions | Delayed Post-intervention Assessment (a 2-month follow up after the completion of the intervention)
  Parents' report of Behavior Rating Inventory of Executive Function, Second Edition (BRIEF2) measuring a range of executive functions, including behavioural, emotional and cognitive regulation

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
The de-identified individual participant data collected during the trial will be available upon reasonable request.
Time Frame: Beginning immediately after publication and ending 5 years after publication.
Access Criteria: To gain access, requestors will need to provide a clear research aim or methodological sound research plan directed to the principal investigator (kkmshum@hku.hk).